CLINICAL TRIAL: NCT06508580
Title: Optimizing Self-Monitoring Feedback Delivery for the Treatment of Obesity
Brief Title: Optimizing Self-Monitoring Feedback for the Treatment of Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202400735
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Micro-randomized 2x2x2x2 factorial model; participants randomized to receive or not receive one of 4 feedback conditions each week for 16 weeks
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Component 1: Calorie Goal Attainment (Experimental): Participants will be randomized to either receive or not receive feedback based on calorie goal attainment.
  Interventions: Behavioral: Component 1: Calorie Goal Attainment
- Component 2: Diet Quality (Experimental): Participants will be randomized to either receive or not receive feedback based on diet quality.
  Interventions: Behavioral: Component 2: Diet Quality
- Component 3: Physical Activity Goal Attainment (Experimental): Participants will be randomized to either receive or not receive feedback based on physical activity goal attainment.
  Interventions: Behavioral: Component 3: Physical Activity Goal Attainment
- Component 4: Goal Setting (Experimental): Participants will be randomized to either receive or not receive feedback based on weekly goal setting.
  Interventions: Behavioral: Component 4: Goal Setting

INTERVENTIONS:
Behavioral: Component 1: Calorie Goal Attainment — On weeks that participants are randomized to receive this component, they will be provided with feedback on the number of days that they met their calorie goal.
  Arms: Component 1: Calorie Goal Attainment
Behavioral: Component 2: Diet Quality — On weeks that participants are randomized to receive this component, they will receive three comments regarding specific dietary choices that may impact weight loss success, including reinforcing comments for behaviors consistent with weight loss and potential areas for change.
  Arms: Component 2: Diet Quality
Behavioral: Component 3: Physical Activity Goal Attainment — On weeks that participants are randomized to receive this component, they will receive feedback related to attainment of that week's physical activity goal.
  Arms: Component 3: Physical Activity Goal Attainment
Behavioral: Component 4: Goal Setting — On weeks that participants are randomized to receive the goal setting component, they will be asked to complete an open-text prompt encouraging them to set a specific weight-related behavior change goal for the next week.
  Arms: Component 4: Goal Setting

SUMMARY:
Self-monitoring (of weight, intake, and activity) is a core component in evidence-based lifestyle interventions for obesity. Research has shown that interventionist feedback increases adherence to self-monitoring and improves weight loss outcomes; however, little empirical evidence exists on how this feedback should be provided. This research study aims to optimize the provision of self-monitoring feedback.

DETAILED DESCRIPTION:
Self-monitoring (e.g., of weight, dietary intake, and physical activity) is a core component in evidence-based comprehensive lifestyle interventions for obesity, and greater adherence to self-monitoring has been associated both with better short-term weight loss and long-term weight loss maintenance. Importantly, research has demonstrated that the provision of interventionist feedback on self-monitoring increases adherence to self-monitoring and improves weight loss outcomes. Little empirical evidence exists, however, to provide guidance on how this feedback should be provided. One study conducted in this area demonstrated that intentions to self-monitor differ by feedback complexity, such that too little (and, conversely, too much) feedback reduces future intentions to self-monitor and engage in related health behavior change; however, less is known regarding how the type and complexity of feedback messages affect actual self-monitoring behavior and subsequent weight loss outcomes. Importantly, provision of this feedback also represents a substantial investment of clinician time; research demonstrated that feedback messages incorporating self-monitoring data related to weight, dietary intake, and physical activity can take ~26 minutes per person to compose. Thus, the investigators propose a line of research that aims to optimize the provision of self-monitoring feedback (i.e., identifying the optimal number and type of feedback messages) for supporting adherence to weight-management behaviors. For the current study, the investigators propose to assess the feasibility and acceptability of a micro-randomized, factorial trial design that will ultimately be used (in a future, fully-powered trial) evaluate the proximal impact of different types and amount of feedback on change in weight and weight-related behaviors (e.g., adherence to self-monitoring, caloric goal attainment, physical activity goal attainment). Using a 2x2x2x2 factorial model, participants will be randomized each week for 16 weeks to one of 16 possible feedback conditions, allowing us to efficiently test four feedback components (i.e., feedback on calorie goal attainment, dietary quality, physical activity goal attainment, or on goal setting) in one study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* BMI ≥ 30.0 kg/m2
* ≤ 175 kg (due to scale limit)
* Own a smartphone (Apple iPhone running iOS 15 or higher or Android smartphone running Android 10 or higher) with a cellular and data plan

Exclusion Criteria:

* Weight > 175 kg (due to a weight limit of the study-provided scale)
* Smartphone device owned deemed incompatible with the Fitbit App
* History of bariatric surgery or plans to obtain bariatric surgery during the study period
* Current use of weight loss medications, or use of weight loss medications in the 6 months prior to initial pre-screening
* Currently participating in a weight-loss program
* Weight loss of ≥ 10 lbs in the 6 months prior to initial pre-screening
* Physical limitations that prevent walking 1/4 mile without stopping
* Use of a pacemaker or other implanted medical device
* Currently pregnant
* Currently breastfeeding
* Less than 1-year post-partum
* Plans to become pregnant within the study period
* Lack of written approval for participation from potential participant's physician if the participant has been diagnosed with diabetes, hypertension, or has a history of coronary heart disease
* One or more study participants living in the household (enrollment limited to one participant per household)
* Medical conditions that contraindicate weight loss or prevent completion of the study (e.g., current diagnosis of cancer or terminal illness, dementia, etc.)
* Self-reported eating disorder within past 5 years
* Unable to complete the 17-week study (due to plans to relocate during the study period, etc.)
* Unable or unwilling to provide informed consent
* Unable to read English at the 5th grade level
* Unwilling to accept random assignment
* Unable or unwilling to download the study smartphone applications, wear the physical activity monitor, or use the study e-scale
* Failure to complete baseline assessment measures
* Failure to complete at least 5 out of 7 days of self-monitoring dietary and weight self-monitoring during the behavioral run-in period
* Other conditions which in the opinion of the Principal Investigator would adversely affect participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Weight | Daily throughout the study period (up to 17 weeks)
  Weight will be assessed using the study-provided e-scales

SECONDARY OUTCOMES:
Frequency of Self-Monitoring Weight | Weekly throughout the study period (up to 17 weeks)
  Frequency of self-monitoring of weight will be defined as the number of days (0-7) each study week that a participant had a valid (e.g., non-outlier) weight recorded via the study-provided e-scale.
Frequency of Self-Monitoring Dietary Intake | Weekly throughout the study period (up to 17 weeks)
  A valid "day" of self-monitoring dietary intake will be defined as ≥ 800 kcal recorded via the Fitbit app or website, consistent with prior research. For each study week, frequency of self-monitoring dietary intake will be defined as the number of valid days (0-7) recorded.
Total Caloric Intake | Weekly throughout the study period (up to 17 weeks)
  For each study week, total caloric intake will be calculated by summing calories recorded via the Fitbit app or website each day of that week between 12:00 AM and 11:59 PM local time.
Calorie Goal Attainment | Weekly throughout the study period (up to 17 weeks)
  Calorie goal attainment each day of the week will be calculated as [TOTAL KCAL INTAKE FOR THE DAY] - [CALORIE GOAL], using calorie data recorded via the Fitbit app or website. Difference scores for the 7 days will be averaged over the week to assess overall adherence to the caloric intake goal during each study week.
Frequency of Self-Monitoring Physical Activity | Weekly throughout the study period (up to 17 weeks)
  Consistent with the broader accelerometry literature, a "valid day" of self-monitoring physical activity will be defined as a day with ≥10 hours of Fitbit wear time, assessed as minutes of non-zero heart rate measurements captured by the Fitbit device. For each study week, frequency of self-monitoring physical activity will be defined as the number of "valid" days (0-7) of Fitbit use.
Physical Activity Minutes | Weekly throughout the study period (up to 17 weeks)
  For each study week, total minutes of physical activity will be calculated by summing the total "active zone minutes" recorded via a Fitbit activity monitor for each day of the week.
Physical Activity Goal Attainment | Weekly throughout the study period (up to 17 weeks)
  For each study week, physical activity goal attainment will be calculated as [TOTAL PHYSICAL ACTIVITY MINUTES] - [PHYSICAL ACTIVITY GOAL], with physical activity minutes recorded via a Fitbit activity monitor.
Feedback Message Acceptability | Weekly throughout the study period (up to 17 weeks)
  Participants will be asked to rate the helpfulness of feedback messages received each week by selecting a "thumbs up" or "thumbs down" button displayed beneath the message.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M Ross, PhD, MPH, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon request following the establishment of an appropriate data use agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The proposed study is a pilot for a larger trial; we will share data from the pilot within one year of completion of the larger trial.